CLINICAL TRIAL: NCT04389008
Title: The Study of Anesthesia-related Risk Factors for Postoperative Death in Elderly Non-cardiac Surgery Patients in China: a Multi-center Retrospective Study Based on Database
Brief Title: The Study of Anesthesia-related Risk Factors for Postoperative Death in Elderly Non-cardiac Surgery Patients in China
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yi Liu, Principal Investigator, Chinese PLA General Hospital
Other Study IDs: PLAGHAOC202001
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Mortality; Anesthesia; Elderly Patients; Noncardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative death
  Interventions: Other: no interventions
- Postoperative non-death
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions

SUMMARY:
At present, the elderly population in China has reached 241 million, and there are more than 20 million elderly surgical patients every year, accounting for about 25% of the surgical population. However, there is no research report on the anesthesia related risk factors of death of elderly patients in hospital. The purpose of this study is to analyze the perioperative data of multicenter database, and to explore the anesthesia related death risk factors of elderly patients with noncardiac surgery in the investigator's country, especially within 24 hours after surgery, so as to help improve the anesthesia management technology of elderly patients during surgery, improve the medical quality of perioperative period, and improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.patients larger than 65 years old at the time of surgery 2.Patients hospitalized for surgery between Jua 2008 to April 2020

Exclusion Criteria:

- 1.Critical demographic information and course records are inaccurate or missing.

2.The outcome could not be determined during the hospitalization. 3.Cardiac surgery patients 4.Patients undergoing surgery under local anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Since January 2008, all the elderly non-cardiac surgery patients have been treated in these four hospitals in the first medical center of PLA general hospital, henan provincial people's hospital, the second xiangya hospital of central south university, the third xiangya hospital of central south university, and the union medical college hospital affiliated to fujian medical university.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2020-05-31 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether death occurred during hospitalization after surgery | Within 30 days after discharge
  Whether death occurred during hospitalization after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No